CLINICAL TRIAL: NCT07011212
Title: In Search of the Correct Diagnosis of Beta-lactam Allergy: From the Validation of a Risk Stratification Tool to Accurate Endotyping
Acronym: Allergy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI24/01913; PI24/01913 (Registry Identifier: Instituto de Salud Carlos III)
Record Dates: First submitted 2025-04-28; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Drug Allergy
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Intervention Model Description: If there are other parties who are masked in the clinical trial besides those listed above, use this space to describe those parties.
Who Masked: Participant
Masking Description: If there are other parties who are masked in the clinical trial besides those listed above, use this space to describe those parties.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL Predictor (Experimental): Parallel,non-inferiority, randomised control trial will be conducted in patients with a low-risk score stratified by BL-Predictor
  Interventions: Diagnostic Test: BL-Predicter
- control (Active Comparator): St followed, if negative,by a fractioned dose DTP wirth 30 min interval between doses: 25%-25%-50% of the maximun dose
  Interventions: Diagnostic Test: BL-Predicter

INTERVENTIONS:
Diagnostic Test: BL-Predicter — To Clinically validate the BL-Predictor toll by a randomised conytrolled ttrial

SUMMARY:
Testing a clinical decision tool (BL-Predictor)

ELIGIBILITY:
Inclusion Criteria:

* signed informed consnet

Exclusion Criteria:

* Use of immunomodulators, antihistamines and corticosteroids

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The main goal of this project is to test a cliniacl decision toll to stratify BL allergic pataients in low and mediaum- anf high-risk | April 2029- june 2027
  And to carry out a deep dissection of the cellular mechanisms of B cells sensitization and basophil and neutrophil activation in BL-IRs to develop accurate in vitro diagnostic test

IPD SHARING:
Plan to Share IPD: No